CLINICAL TRIAL: NCT01864005
Title: A Multicentre, Open-label, Randomized, 6-week, Phase IV Study of the Onset and Maintenance of the Antiplatelet Effect of Ticagrelor Compared With Clopidogrel With Aspirin as Background Therapy in Chinese Patients With Non-ST or ST Elevation Acute Coronary Syndromes (ACS)
Brief Title: A Phase IV Study of the Onset and Maintenance of the Antiplatelet Effect of Ticagrelor Compared With Clopidogrel in Chinese Patients With ACS
Acronym: HouYi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5130L00053
Record Dates: First submitted 2013-05-24; First posted 2013-05-29 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Non-ST or ST Elevation Acute Coronary Syndromes
Keywords: Non-ST or ST Elevation Acute Coronary Syndromes, Ticagrelor, Clopidogrel, Antiplatelet Effect
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental)
  Interventions: Drug: Ticagrelor
- clopidogrel (Active Comparator)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — 90mg tablets. loading dose of 180mg ticagrelor tablets (two 90mg tablets) taken orally, followed by 90mg of ticagrelor 12 hours after the first dose. Duration of treatment: 6 weeks.
  Arms: Ticagrelor
Drug: Clopidogrel — 75mg capsule. loading dose of 600mg clopidogrel capsules (eight 75mg capsules) taken orally, follow by 75mg of clopidogrel capsules orally od. Duration of treatment: 6 weeks.
  Arms: clopidogrel

SUMMARY:
The purpose of this study is to test the hypothesis that the onset of the antiplatelet effect of ticagrelor is more rapid and greater than clopidogrel in Chinese patients with ACS.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provision of informed consent prior to any study specific procedures
* 2. Female or male aged at least 18 years
* 3. Females of child-bearing potential must have a negative urine pregnancy test at enrolment and be willing to use reliable contraception
* 4. Index event of non-ST or ST segment elevation ACS.

Exclusion Criteria:

* 1.Contraindication or other reason that clopidogrel or ticagrelor should not be administered (eg, hypersensitivity, active bleeding, moderate or severe liver disease, history of previous intracranial bleed, GI bleed within the past 6 months, major surgery within 30 days)
* 2. Oral anticoagulation therapy or GP IIb/IIIa receptor antagonists therapy within 30 days prior to randomisation or cannot be stopped
* 3. Ticagrelor or clopidogrel or other P2Y12 inhibitors within 14 days prior to randomisation
* 4. Requires dialysis
* 5. Nonselective non-steroidal anti-inflammatory drugs (NSAIDs) and prostacyclins (PGI2) therapy that cannot be stopped

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, Professor, Principal Investigator — The General Hospital of People's Liberation Army
Locations (3):
- China (3):
  - Research Site, Beijing
  - Research Site, Shenyang
  - Research Site, Tianjin

REFERENCES:
- See also: D5130L00053_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1828&filename=D5130L00053_CSR_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 15/05/2013, Last subject last visit: 18/03/2014. There were 5 study centers in China, which participated this study.
Pre-assignment Details: There was no run-in or any other pre-assignment periods following participant enrollment.
Groups:
- Ticagrelor: Patients received a loading dose of 180mg ticagrelor tablets (two 90mg tablets) taken orally, followed by 90mg of ticagrelor 12 hours after the first dose. The third dose of ticagrelor was given to patients after the blood sample had been obtained 24 hours after the first dose. Thereafter, the patients took 90mg of ticagrelor orally bd. The total study period was 6 weeks.
- Clopidogrel: Patients received a loading dose of 600mg clopidogrel tablets (eight 75mg tablets) taken orally. The second dose of clopidogrel had been given to patients after the blood sample had been obtained 24 hours after the first dose. Thereafter, the patients took 75mg of clopidogrel orally od. The total study period was 6 weeks.
Period: Overall Study
Arm/Group | Ticagrelor | Clopidogrel
Started | 29 | 31
Completed | 26 | 25
Not Completed | 3 | 6
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Incorrect enrolment | 1 | 0
Not completed — Disease need | 1 | 1
Not completed — Need GP IIb/IIIa | 1 | 3

BASELINE CHARACTERISTICS:
Population: Three randomized patients were excluded from the full analysis set (FAS) due to any of the following reasons: 1) did not meet exclusion requirments but was randomized, 2)post-treatment blood PRU was not available, 3) pre-treatment blood PRU was missing, and 4) use of prohibited medications.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor | Clopidogrel | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.75 (10.967) | 58.59 (9.789) | 58.67 (10.291)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 10
  Male | 26 | 21 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 28 | 29 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: the Percentage Inhibition of the P2Y12 Receptor
Description: Note: the primary endpoint was changed per the statistical analysis plan prior database lock.
Time Frame: at 2 hours after first dose of study drug
Population: FAS (full analysis set). Three randomized patients were excluded from FAS due to any of the following reasons: 1) did not meet exclusion requirments but was randomized, 2)post-treatment blood PRU was not available, 3) pre-treatment blood PRU was missing, and 4) use of prohibited medications.
Measure: Mean (Standard Deviation); unit: Percentage Inhibition
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 28 | 29
Percentage Inhibition | 48.20 (45.410) | 9.78 (27.574)
Statistical Analysis 1: Comparison: Ticagrelor vs Clopidogrel; Test type: Superiority or Other; p = 0.0021, Wilcoxon (Mann-Whitney) — not adjusted for multiple comparisons. statistical significance level: 0.05
Statistical Analysis 2: Comparison: Ticagrelor vs Clopidogrel; Test type: Superiority or Other; p = 0.0003, ANOVA; Mean Difference (Final Values) = 38.421, 95% CI 2-sided [18.559 to 58.283]

2. Secondary Outcome: the Percentage Inhibition of the P2Y12 Receptor
Time Frame: at 0.5 hour after first dose of study drug
Population: PPS (per-protocol set). Seven randomized patients were excluded from PPS due to any of the following reasons: 1) did not meet exclusion requirments but was randomized, 2)post-treatment blood PRU was not available, 3) pre-treatment blood PRU was missing, 4) missing blood PRU at 2h after first dose, and 5) use of prohibited medications.
Measure: Mean (Standard Deviation); unit: Percentage Inhibition
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 26 | 27
Percentage Inhibition | 8.23 (25.810) | -3.91 (13.602)
Statistical Analysis 1: Comparison: Ticagrelor vs Clopidogrel; Test type: Superiority or Other; p = 0.0828, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: the Percentage Inhibition of the P2Y12 Receptor
Time Frame: at 8 hours after first dose of study drug
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage Inhibition
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 26 | 27
Percentage Inhibition | 67.91 (34.856) | 25.38 (32.738)
Statistical Analysis 1: Comparison: Ticagrelor vs Clopidogrel; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: the Percentage Inhibition of the P2Y12 Receptor
Time Frame: at 24 hours after first dose of study drug
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage Inhibition
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 26 | 27
Percentage Inhibition | 79.25 (17.920) | 28.76 (26.917)
Statistical Analysis 1: Comparison: Ticagrelor vs Clopidogrel; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: the Percentage Inhibition of the P2Y12 Receptor
Time Frame: at 6 weeks after first dose of study drug
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage Inhibition
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 26 | 27
Percentage Inhibition | 83.78 (13.947) | 24.22 (33.546)
Statistical Analysis 1: Comparison: Ticagrelor vs Clopidogrel; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 weeks for all AEs and another 14 days for SAEs.
Arm/Group | Ticagrelor | Clopidogrel
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/31
Other Adverse Events (participants affected / at risk) | 12/29 | 12/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=29) | Clopidogrel (N=31)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ticagrelor (N=29) | Clopidogrel (N=31)
Hypertensive heart disease (Cardiac disorders) | 3 | 2
Arrhythmia (Cardiac disorders) | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Puncture site infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Blood creatine increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
(1) Sample size was relatively small. (2) Study duration with 6 weeks seemed limited. (3) Sampling time-points seemed relatively scarce, such as missing the time point for 1-hour and 4-hour after loading dose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days